CLINICAL TRIAL: NCT06839742
Title: Does the Addition of a Deep Posterior Gluteal Compartment Block to Suprainguinal Fascia Iliaca Block Improve Analgesia in Hip Fracture Surgery? A Randomized Controlled Trial
Brief Title: Does Adding Posterior Block to SFIB Increase the Quality of Analgesia in Hip Fractures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OMUKAEAK 2024/276
Record Dates: First submitted 2024-12-11; First posted 2025-02-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Acute Pain Management; Hip Surgery
Keywords: acute pain management; hip surgery; Deep posterior gluteal compartment block; Suprainguinal fascia iliaca plane block

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SFICB (Active Comparator): Suprainguinal fascia iliaca plane block will be performed 30 minutes before hip surgery
  Interventions: Other: Suprainguinal fascia iliaca compartment block
- Group Combined (Active Comparator): Suprainguinal Fascia İliaca plane Block will be performed 30 minutes before hip surgery and Deep Posterior Gluteal Compartment Block will be performed 20 minutes before hip surgery
  Interventions: Other: Deep Posterior Gluteal Compartment Block; Other: Suprainguinal fascia iliaca compartment block

INTERVENTIONS:
Other: Deep Posterior Gluteal Compartment Block — Deep Posterior Gluteal Compartment Block will be performed under USG guidance before neuraxial anesthesia.
  Arms: Group Combined
Other: Suprainguinal fascia iliaca compartment block — Suprainguinal fascia iliaca compartment block will be performed under USG guidance before neuraxial anesthesia.

SUMMARY:
The researchers aimed to compare the effects of adding a Deep Posterior Gluteal Compartment Block to a Suprainguinal Fascia Iliaca Compartment Block (SFICB) versus SFICB alone on pain, analgesic consumption, and positioning pain for neuraxial anesthesia.

DETAILED DESCRIPTION:
Adding Deep Posterior Gluteal Compartment Block to Suprainguinal Fascia Iliaca Block applied before neuraxial anesthesia in hip fracture surgeries can reduce the pain sensation originating from the posterior region of the hip joint. Thus, participants can experience less pain in the perioperative period, consume less analgesics and reduce complications related to these in the postoperative period. In addition, possible complications can be prevented with early mobilization of the participants. It was aimed to compare the effects of adding Deep Posterior Gluteal Compartment Block to Suprainguinal Fascia Iliaca Block with only Suprainguinal Fascia Iliaca Block on these results.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Patients between the ages of 18-90
* ASA I, II, III
* Patients whose surgery duration does not exceed 2 hours
* Patients who will undergo surgery under spinal anesthesia

Exclusion Criteria:

* Patients who do not want to participate in the study/do not give consent
* Patients with a condition that prevents regional anesthesia
* Patients with cognitive dysfunction who are unable to evaluate the NRS score and who cannot use PCA (Patient Controlled Analgesia Device)
* History of hypersensitivity or allergy to local anesthetics
* Patients with psychiatric disorders and those using psychiatric medications
* Presence of hematological disease
* Presence of oncological disease
* Patients with serious major organ failure
* Presence of multiple fractures
* Patients with alcohol or drug addiction
* Patients who have used analgesic drugs up to 12 hours before surgery
* ASA IV-V patients
* Morbidly obese patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours
  In the postoperative period, patients will be given opioids according to their pain density with a patient-controlled device, and the daily Morphine consumption in Patient Controlled Analgesia device will be collected and compared between groups.

SECONDARY OUTCOMES:
Perioperative pain intensity | 24 hours
  Changes in the Numerical Rating Scale (NRS) will be recorded at rest and during movement. The participant's baseline NRS will be recorded, followed by measurements before and after neuraxial positioning and up to 24 hours post-surgery.
  The NRS is a unidimensional measure of pain intensity in adults. It is a segmented numerical version of the Visual Analog Scale (VAS) where the participant selects a whole number (0-10) that best represents the intensity of their pain. The 11-point numerical scale ranges from '0' representing one end of the pain spectrum (e.g. 'no pain') to '10' representing the other end (e.g. 'worst imaginable pain').
Quality of recovery 15 scale | 24 hours after surgery
  Postoperative Quality of Recovery 15 in Turkish scale
Quality of patient's position for neuraxial anesthesia | up to ten minutes
  The position will be evaluated by anesthesiologist and characterized as "unsatisfactory", "satisfactory", "good" or "very good"
Quadriceps weakness | 24th hours
  Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE SELÇUK KUŞDERCİ, Study Director — SAMSUN UNİVERSITY
Locations (1):
- Samsun University, Samsun Training and Research Hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Safa B, Trinh H, Lansdown A, McHardy PG, Gollish J, Kiss A, Kaustov L, Choi S. Ultrasound-guided suprainguinal fascia iliaca compartment block and early postoperative analgesia after total hip arthroplasty: a randomised controlled trial. Br J Anaesth. 2024 Jul;133(1):146-151. doi: 10.1016/j.bja.2024.04.019. Epub 2024 May 18. PMID 38762396
- [Background] Roche JJ, Wenn RT, Sahota O, Moran CG. Effect of comorbidities and postoperative complications on mortality after hip fracture in elderly people: prospective observational cohort study. BMJ. 2005 Dec 10;331(7529):1374. doi: 10.1136/bmj.38643.663843.55. Epub 2005 Nov 18. PMID 16299013
- [Background] Vermeylen K, Van Aken D, Versyck B, Casaer S, Bleys R, Bracke P, Groen G. Deep posterior gluteal compartment block for regional anaesthesia of the posterior hip: a proof-of-concept pilot study. BJA Open. 2023 Feb 15;5:100127. doi: 10.1016/j.bjao.2023.100127. eCollection 2023 Mar. PMID 37587997